CLINICAL TRIAL: NCT02456532
Title: Risks for Transition From Therapeutic Hypnotic Use to Abuse
Brief Title: Safety and Efficacy of Chronic Hypnotic Use 2
Acronym: CIS2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Timothy Roehrs, PhD, Senior Bioscientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #9384
Record Dates: First submitted 2015-05-06; First posted 2015-05-28 (Estimated); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-07

CONDITIONS: Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Intervention: Six months of nightly placebo
  Interventions: Drug: placebo
- Zolpidem CR (Active Comparator): Intervention: Six months of zolpidem cr 12.5 mg nightly use
  Interventions: Drug: Zolpidem CR
- Eszopiclone (Active Comparator): Intervention: Six months of eszopiclone 3 mg nightly use
  Interventions: Drug: Eszopiclone

INTERVENTIONS:
Drug: placebo — six months of nightly placebo
  Arms: Placebo
Drug: Zolpidem CR — six months of nightly zolpidem
  Other Names: Ambian CR
  Arms: Zolpidem CR
Drug: Eszopiclone
  Other Names: Lunesta
  Arms: Eszopiclone

SUMMARY:
This proposal will assess risks for transition from therapeutic hypnotic use to abuse in people with insomnia. The investigators will study a hypothesized at-risk sub-population, insomniacs with hyperarousal, and compare two hypnotics, a drug with mood effects, eszopiclone, versus one without mood effects, zolpidem.

DETAILED DESCRIPTION:
Persons with DSM-V diagnosed insomnia disorder, aged 18-65 yrs, with no other sleep disorders, unstable medical or psychiatric diseases or drug dependency will be entered to the trial. Following a screening NPSG and MSLT, participants will be randomized to zolpidem XR 12.5 mg (n=60), eszopiclone 3 mg (n=60), or placebo (n=50) nightly for 6 months. After 6 months of nightly use, over a 2-week choice period, they were instructed to discontinue hypnotic use, but if necessary, to self-administer either 1, 2, or 3 capsules of their assigned "blinded" medication (zolpidem XR 6.25 mg, 6.25 mg, placebo; eszopiclone 2 mg, 1 mg, placebo as capsules 1, 2 and 3 respectively; or 3 placebos). Nightly sleep at home will be recorded by actigraphy for one week after the screening NPSG and MSLT and before treatment is initiated and actigraphy again during the two week discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of insomnia

Exclusion Criteria:

* acute or unstable medical disease,
* current or past history of psychiatric disease, alcoholism or drug abuse, and other primary sleep disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Roehrs, PhD, Principal Investigator — Henry Ford Health System Sleep Disorders Ctr
Locations (1):
- HFHS Sleep Disorders Ctr, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Intervention: Six months of nightly placebo
  placebo
- Zolpidem CR: Intervention: Six months of zolpidem cr 12.5 mg nightly use
  Zolpidem CR
- Eszopiclone: Intervention: Six months of eszopiclone 3 mg nightly use
  Eszopiclone
Period: Overall Study
Arm/Group | Placebo | Zolpidem CR | Eszopiclone
Started | 14 | 11 | 16
Completed | 14 | 11 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Zolpidem CR | Eszopiclone | Total
Number analyzed (Participants) | 14 | 11 | 16 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 16 | 41
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (9.1) | 42.5 (10.8) | 41.1 (12.6) | 43.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 14 | 36
  Male | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Count of Participants: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Count of Participants: Asian | 2 | 1 | 0 | 3
  Count of Participants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Count of Participants: Black or African American | 8 | 3 | 8 | 19
  Count of Participants: White | 4 | 7 | 8 | 19
  Count of Participants: More than one race | 0 | 0 | 0 | 0
  Count of Participants: Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 16 | 41
Baseline PSG defined sleep efficiency [Mean (Standard Deviation); unit: percent sleep per 8 hrs] | 75.2 (15.9) | 75.7 (10.5) | 78.7 (13.0) | 76.7 (13.3)
Average daytime sleep latency in min [Mean (Standard Deviation); unit: minutes] | 11.1 (5.1) | 11.9 (6.5) | 11.7 (5.1) | 11.5 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Capsules Taken During Discontinuation From Either Active Drug vs Placebo Over a Two Week Period
Description: instruction to stop nightly hypnotic use over a two-week discontinuation period with option to choose of 1, 2, 3 capsules, if necessary
Time Frame: total number of capsules chosen in week 1 and week 2 of the discontinuation period
Measure: Mean (Standard Deviation); unit: Total number capsules chosen
Arm/Group | Placebo | Zolpidem CR | Eszopiclone
Number analyzed (Participants) | 14 | 11 | 16
Total number capsules chosen | 0.43 (1.6) | 2.6 (4.5) | 6.3 (10.5)
Statistical Analysis 1: Comparison: Placebo vs Zolpidem CR vs Eszopiclone; Test type: Other — analyses of variance comparing the three treatment gropus; p = 0.05, ANOVA

2. Secondary Outcome: Percent of Time Asleep Over Time in Bed During the Two-week Discontinuation Period
Description: comparing the three treatment arms for nightly hypnotic efficacy using actigraphic determined sleep efficiency over the two week discontinuation period
Time Frame: mean nightly sleep efficiency during week 1 and week 2 of the discontinuation period
Measure: Mean (Standard Deviation); unit: % sleep time/bedtime
Arm/Group | Placebo | Zolpidem CR | Eszopiclone
Number analyzed (Participants) | 14 | 11 | 16
% sleep time/bedtime | 81.9 (8.1) | 84.4 (5.1) | 83.0 (4.9)
Statistical Analysis 1: Comparison: Placebo vs Zolpidem CR vs Eszopiclone; Test type: Other — ANOVA; p = 0.643, ANOVA

ADVERSE EVENTS:
Time Frame: 6 months
Description: reported weekly by questionnaire
Arm/Group | Placebo | Zolpidem CR | Eszopiclone
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11 | 0/16

LIMITATIONS AND CAVEATS:
Difficulty reaching proposed enrollment target: 41 of projected 120 participants completed the study- in part due to COVID. Study is to be considered preliminary

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT02456532/Prot_SAP_000.pdf